CLINICAL TRIAL: NCT06231147
Title: Effects of Horse Riding Simulator With or Without Visual Feedback on Balance and Postural Control in Children With Spastic Cerebral Palsy
Brief Title: Effects of Horse Riding Simulator With or Without Visual Feedback on Balance and Postural Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: REC/RCR&AHS/23/0765
Record Dates: First submitted 2023-12-26; First posted 2024-01-30 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy
Keywords: Balance; Cerebral Palsy; Horse Riding Simulator (HRS); Posture Control
MeSH Terms: conditions — Cerebral Palsy | interventions — Feedback, Sensory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): horse riding simulator sessions with mirror visual feedback
  Interventions: Other: HORSE RIDING SIMULATOR WITH VISUAL FEEDBACK
- Group B (Other): horse riding simulator sessions without mirror visual feedback
  Interventions: Other: HORSE RIDING SIMULATOR WITHOUT VISUAL FEEDBACK

INTERVENTIONS:
Other: HORSE RIDING SIMULATOR WITH VISUAL FEEDBACK — horse riding simulator session with mirror visual feedback. The participants will be instructed that how to perform exercises by using the horse riding simulator (HRS) system in front of mirror
  Arms: Group A
Other: HORSE RIDING SIMULATOR WITHOUT VISUAL FEEDBACK — horse riding simulator session without visual feedback. The participants will be instructed that how to perform exercises by using the horse riding simulator (HRS) system.
  Arms: Group B

SUMMARY:
Spastic cerebral palsy is a neurological condition that causes muscle spasticity and motor impairments, greatly impacting a child's ability to maintain balance and control their posture. The horse riding simulator (HRS), inspired by hippo therapy, has emerged as a potential therapeutic intervention for enhancing motor function in individuals with cerebral palsy. This study explored the additional effects of mirror visual feedback when used in conjunction with the HRS. Strategically placed mirrors allow participants to observe their own body movements and positions in real-time. The simulator's rhythmic, multidimensional movements deliver sensory input and challenge the motor system, promoting postural adjustments and improved balance. Furthermore, the integration of mirror visual feedback appears to enhance the therapeutic benefits. Real-time visual information enables children to actively observe and correct their body positioning, leading to improved body awareness and more efficient motor responses.

DETAILED DESCRIPTION:
Cerebral palsy (CP), one of the most common physical disabilities in childhood, is a disorder of movement and posture caused by non-progressive lesions in the developing brain. Children with CP, to varying degrees, have muscle weakness, tone abnormality, and motor-control impairment, causing abnormal posture and poor balance control.In high-income countries, the current birth prevalence of cerebral palsy has decreased to 1.6 per 1000 live births. However, in low- and middle-income countries, the birth prevalence is significantly higher. Children diagnosed with CP exhibit a range of muscle weakness, tone abnormalities, and impaired motor control. These factors contribute to abnormal posture and compromised control over balance

ELIGIBILITY:
Inclusion Criteria:

* Spastic cerebral palsy with level I and II according to Gross Motor Function Classification System (GMFCS)
* Age between 8 and 12 years
* Ability to sit and stand independently
* Both genders are included (female and male)

Exclusion Criteria:

* Having received an injection of botulinum toxin within 3 months
* Having undergone orthopedic surgery or selective dorsal rhizotomy in the previous 1 year
* Having undergone HRS training within 6 months;
* Having severe pain, joint dislocation, contracture, or spinal deformity
* Having experienced uncontrolled epileptic seizure
* Having poor visual or hearing acuity.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Pediatric balance scale | 8 weeks
  The Pediatric Balance Scale is assessment tool specifically designed to evaluate balance in children. It has been extensively used in clinical and research settings to assess balance impairments and monitor progress over time.
Posture and postural ability scale | 8 weeks
  Posture and Postural Ability Scale is an assessment tool that allows for posture and postural ability to be assessed independently

CONTACTS AND LOCATIONS:
Overall Officials: Shehar Bano, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jung YG, Chang HJ, Jo ES, Kim DH. The Effect of a Horse-Riding Simulator with Virtual Reality on Gross Motor Function and Body Composition of Children with Cerebral Palsy: Preliminary Study. Sensors (Basel). 2022 Apr 10;22(8):2903. doi: 10.3390/s22082903. PMID 35458888